CLINICAL TRIAL: NCT06578481
Title: The Effect of Postural Stabilization Exercises on Craniovertebral Angle, Disability and Quality of Life in Patients With Chronic Neck Pain: Randomized Controlled Trial
Brief Title: The Effectiveness of Postural Stabilization Exercises in Patients With Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European University of Lefke (Other)
Responsible Party: Principal Investigator, Gölgem Mehmetoğlu, Lecturer, European University of Lefke
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EULefke
Record Dates: First submitted 2024-08-26; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SLPS Group (Experimental): Scapular and lumbopelvic stabilization group
  Interventions: Other: Exercises
- CS group (Active Comparator): Cervical stabilization group
  Interventions: Other: Exercises

INTERVENTIONS:
Other: Exercises — Individuals in the first group underwent cervical stabilization (CS) exercises and additional scapular and lumbopelvic stabilization (SLPS) exercises three times a week for 6 weeks. The second group was treated with only CS exercises for the same period. In addition, stretching exercises and a 20-minute hot pack were applied to the muscles around the neck of all patients.

SUMMARY:
This study aimed to evaluate the effect of postural stabilization exercises given in addition to cervical stabilization on craniovertebral angle, neck disability index, and quality of life in people with chronic neck pain.Sixty women with chronic neck pain between the ages of 20-60 were included in the study and the individuals were randomly divided into two groups. Individuals in the first group underwent cervical stabilization (CS) exercises and additional scapular and lumbopelvic stabilization (SLPS) exercises three times a week for 6 weeks. The second group was treated with only CS exercises for the same period. In addition, stretching exercises and a 20-minute hot pack were applied to the muscles around the neck of all patients. Craniovertebral angle (CVA) was measured by photogrammetry. Disability level was measured by the Neck Disability Index (NDI). The Turkish version of the Short Form-36 (SF-36) was used to assess quality of life.

ELIGIBILITY:
Inclusion Criteria:

* The study included females between the ages of 20-60 years, with moderate pain intensity (3 cm and above according to the Visual Pain Scale) and neck pain lasting more than 3 months.

Exclusion Criteria:

* Participants who had undergone any shoulder or neck surgery complained of fibromyalgia and myofascial pain syndrome, had a neurological disease, cervical radiculopathy, and serious systemic disease that would interfere with treatment, and who were pregnant were excluded from the study

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Craniovertebral Angle Measurement | 6 weeks
  The craniovertebral angle (CVA) is formed by the intersection of a horizontal line passing through the seventh cervical vertebra in the sagittal plane and a line going to the tragus of the ear
Neck Disability Index | 6 weeks
  The Neck Disability Index was used to assess the disability of people with chronic neck pain during daily activities
Health Related Quality of Life | 6 weeks
  The Turkish version of the Short Form-36 (SF-36) is used to assess health-related quality of life. Short Form-36 (SF-36) is a self-assessment scale and analyses 8 dimensions of health

CONTACTS AND LOCATIONS:
Locations (1):
- European University of Lefke, Lefka, Gemikonağı, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mehmetoglu G, Yuksel I. Effect of Postural Stabilization Exercises in Combination with Cervical Stabilization Exercises on Craniovertebral Angle, Pain, Disability, and Quality of Life in Patients with Chronic Neck Pain: A Randomized Controlled Trial. Healthcare (Basel). 2025 Jun 11;13(12):1388. doi: 10.3390/healthcare13121388. PMID 40565415